CLINICAL TRIAL: NCT06493513
Title: The Effect of 40 Hz Transcranial Stimulation on the Incidence of Emergence Delirium After Sevoflurane Anesthesia in Children
Brief Title: The Effect of 40 Hz Transcranial Stimulation on the Incidence of Emergence Delirium in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Henan-FSH
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Emergence Delirium; Anesthesia; Children
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Experimental group: at the onset of anesthesia, the child received 40Hz transcranial stimulation for 1h.
  Control group: at the start of anesthesia, the child did not receive any additional treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized (like flipping a coin or drawing from a hat) to either of the two groups, with the probability of a participant being in the experimental and control groups being 1:1. and neither participant, nor care Provider, nor the outcome assessor, nor the investigator will know to which group participant has been assigned (or add 40 Hz transcranial stimulation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 40Hz stimulation group (Experimental): At the start of anesthesia, the child received 40Hz transcranial stimulation for 1h.
  Interventions: Device: 40Hz stimulation
- Control group (No Intervention): At the start of anesthesia, the child did not receive any additional treatment.

INTERVENTIONS:
Device: 40Hz stimulation — Exogenous 40Hz stimulation is a physical intervention that induces gamma oscillations, oscillations and pulsations at the corresponding frequency, and may lead to a significant reduction in β-amyloid, reversal of tau protein hyperphosphorylation, and consequently improvement of cognitive function in patients.
  Arms: 40Hz stimulation group

SUMMARY:
Emergence delirium is a complex of perceptual deficits and psychomotor agitation most commonly seen in preschool children in the early post-anesthetic period. It increases the risk of bed falls, accidental catheter removal, surgical wound dehiscence, and delayed discharge in children. Exogenous 40 Hz stimulation can improve cognitive functioning. Therefore, the aim of this study was to explore the effect of 40Hz stimulation on the incidence of emergence delirium in children undergoing vascular malformation surgery under sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-14 years old
2. ASA classification I or II
3. Proposed vascular malformation surgery under sevoflurane general anesthesia
4. Anesthesia duration>1h
5. Obtaining informed consent

Exclusion Criteria:

1. Emergency surgery
2. Mental retardation
3. Neurological disorders with manic-like symptoms
4. Presence of severe kidney or liver disease, heart or respiratory disease
5. Autoimmune diseases
6. Vascular malformation of the head and face
7. Significant life changes in the 1 month prior to surgery

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence delirium | From extubation to 2 h after extubation and day 1, day 2, day 3 after surgery.
  Emergence delirium was considered to have occurred in the subject child if Pediatric Anesthesia Emergence Delirium (PAED) scale ≥10 or Cornell Assessment of Pediatric Delirium (CAPD) scale ≥10 (PAED range: 0-20 points, CAPD range: 0 ~ 32 points).

SECONDARY OUTCOMES:
The incidence of pain | Day 1, day 2, day 3 after surgery.
  If the Face, Legs, Activity, Cry and Consolability (FLACC) scale ≥ 4 (0 [no pain] ~ 10 [worst pain]), the child was considered to be in pain.
The incidence of postoperative nausea and vomiting | Day 1, day 2, day 3 after surgery.
  Follow up patients for nausea and vomiting
Sleep quality | Day 1, day 2, day 3 after surgery.
  Assessment of children's daily sleep quality by Self-Rating Scale of Sleep (SRSS), with a score range of 10 ~ 50, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu S, Bian J, Fu Y, Yang Y, Wang Y, Zhu G, Ruan X, Li N, Wang D, Zhang J, Sun M. 40-Hz Light Stimulation and Emergence Delirium Incidence After Sevoflurane Anesthesia in Children: A Randomized Clinical Trial. JAMA Pediatr. 2025 Dec 1;179(12):1300-1307. doi: 10.1001/jamapediatrics.2025.3903. PMID 41082242